CLINICAL TRIAL: NCT04250493
Title: Insulin Resistance in Multiple System Atrophy
Acronym: IRAMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: University of Bordeaux (Other); Labex Brain (Other); Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CHUBX 2018/30
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Multiple System Atrophy
Keywords: Multiple system atrophy; Neurodegenerative disease; Alpha synuclein; Insulin resistance
MeSH Terms: conditions — Multiple System Atrophy; Neurodegenerative Diseases; Parkinson Disease 4, Autosomal Dominant Lewy Body; Insulin Resistance | interventions — Mental Status and Dementia Tests; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSA patient (Experimental): Patients will be recruited at the French Reference Center for MSA.
  Interventions: Biological: Homeostasis Model Assessment of insulin resistance (HOMA); Behavioral: MOntreal Cognitive Assessment (MoCA); Behavioral: Clinical characteristics of AMS patients; Procedure: Brain Magnetic Resonance Imaging (MRI); Biological: Blood sampling
- Control (Other): Healthy volunteer matched for age (+/- 5years) and sex with MSA patient.
  Interventions: Biological: Homeostasis Model Assessment of insulin resistance (HOMA); Behavioral: MOntreal Cognitive Assessment (MoCA); Procedure: Brain Magnetic Resonance Imaging (MRI); Biological: Blood sampling

INTERVENTIONS:
Biological: Homeostasis Model Assessment of insulin resistance (HOMA) — Fasting blood sample for : glucose, insulinemia, hemoglobin and lipid test to determine the Homeostasis Model Assessment of insulin resistance (HOMA) index
Behavioral: MOntreal Cognitive Assessment (MoCA) — Cognitive evaluation with MOntreal Cognitive Assessment (MoCA)
Behavioral: Clinical characteristics of AMS patients — Severity and progression of motor disorders assessed by the UMSARS scale, severity of dysautonomia assessed by the COMPASS31 scale ; quality of life questionnaire (AMS-Qol) for the level of difficulty experienced by the patient (on activities such as : move; walk; maintain balance; talk; feed)
  Arms: MSA patient
Procedure: Brain Magnetic Resonance Imaging (MRI) — Brain Magnetic Resonance Imaging (MRI) : putamen imaging, bridge and cerebellum; white substance hypersignals volume
Biological: Blood sampling — Optional blood sampling for the constitution of a biological collection

SUMMARY:
Multiple system atrophy (MSA) is a rare and fatal neurodegenerative disorder. The pathologic hallmark is the accumulation of aggregated alpha-synuclein in oligodendrocytes forming glial cytoplasmic inclusions. Some symptomatic treatments are available while disease-modification remains an unmet treatment need. Post-mortem findings suggest insulin resistance, i.e. reduced insulin signaling, in the brains of MSA patients. The aim of this study is to complete the target validation of insulin resistance for future treatment trials.

DETAILED DESCRIPTION:
Multiple system atrophy (MSA) patients have a poor prognosis with a median survival ranging between 6 and 10 years. MSA belongs to the synucleinopathies, which are characterized by the abnormal accumulation of alpha-synuclein. We have recently shown brain insulin resistance (i.e. reduced insulin signaling) in post-mortem brain tissue of MSA patients and transgenic MSA mice, as illustrated by increased protein levels of insulin receptor substrate-1 phosphorylated at serine 312 (IRS-1pS312). Additionally, exendin-4, an approved anti-diabetic drug targeting glucagon-like peptide-1 (GLP-1) receptors, was capable of decreasing brain levels of IRS-1pS312 and preserving dopamine neurons in transgenic MSA mice. We further observed an inverse correlation between plasma neural-derived exosomal IRS-1pS312 levels and survival of dopamine neurons in transgenic MSA mice.

The aim of this study is to further characterize peripheral and central insulin resistance in MSA patients, thereby validating this target for future treatment trials. For this purpose, fasting blood glucose and insulin levels will be determined in samples of MSA patients and healthy controls for a homeostatic model assessment of insulin resistance (HOMA). Additionally, IRS-1pS312 will be measured in neural-derived plasma exosomes of MSA patients and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

Patients :

* Patients suffering from "possible" or "probable" MSA according to clinical consensus criteria (Gilman et al., 2008).
* Age > 30
* Written informed consent
* Patient covered by the national health system

Controls:

* Patients not suffering from a neurologic disorder
* Age > 30
* Written informed consent
* Patient covered by the national health system

Exclusion Criteria:

For patients and controls:

* Presence of a diabetes
* Treatment with corticosteroids, estrogen, atypical antipsychotics, and anti-retroviral agents
* Patient under tutelage
* Patient unable to give consent
* Any other neurologic disorder
* Pregnancy and breastfeeding
* MOCA ≤21
* Contraindication to perform an MRI

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2020-10-28 (Actual); Primary Completion 2026-10-28 (Estimated); Study Completion 2027-10-28 (Estimated)

PRIMARY OUTCOMES:
HOMA Index | Day 0
  Homeostasis Model Assessment of insulin resistance (HOMA) index, calculated from a fasted blood glucose and insulin level between AMS patients and a formula-controlled group (insulinemia x glycemia)/22.5 insulinemia being expressed in mU/l and glucose in mmol/L.

SECONDARY OUTCOMES:
IRS-1pS312 (Insulin Receptor Substrate-1, Phosphorylated at Serine 312) concentration | Day 0
  Mean concentration of neuronal IRS-1pS312 in plasma exosomes
Unified Multiple System Atrophy Rating Scale (UMSARS) score | Day 0
  UMSARS I (0=no disorder, 48=severe disorders): is an evaluation of activities of daily life via 12 items. It evaluates language, writing, autonomy (diet; dressing; hygiene), walking and the presence of possible urinary, sexual or intestinal disorders.
  UMSARS II (0=no disorder, 56=severe disorders): consists of a motor examination on the basis of 14 items that allow to evaluate including facial expression, oculomotricity, oral expression, tremors or walking.
  UMSARS III: consists of measurements of blood pressure and heart rate in the lying and standing position for 10 minutes every minute.
  UMSARS IV : disability assessment from 1 to 5 (1= completely independent; 5 = totally dependent / dependent)
Unified Multiple System Atrophy Rating Scale (UMSARS) score | One year
  UMSARS I (0=no disorder, 48=severe disorders): is an evaluation of activities of daily life via 12 items. It evaluates language, writing, autonomy (diet; dressing; hygiene), walking and the presence of possible urinary, sexual or intestinal disorders.
  UMSARS II (0=no disorder, 56=severe disorders): consists of a motor examination on the basis of 14 items that allow to evaluate including facial expression, oculomotricity, oral expression, tremors or walking.
  UMSARS III: consists of measurements of blood pressure and heart rate in the lying and standing position for 10 minutes every minute.
  UMSARS IV : disability assessment from 1 to 5 (1= completely independent; 5 = totally dependent / dependent)
COMPosite Autonomic Symptoms Score (COMPASS-31) | Day 0
  Assessment of dysautonomia. The scale consists of 31 items in 6 domains and provides an autonomic symptom score from 0 to 100. High values represent severe symptoms
COMPosite Autonomic Symptoms Score (COMPASS-31) | One year
  Assessment of dysautonomia. The scale consists of 31 items in 6 domains and provides an autonomic symptom score from 0 to 100. High values represent severe symptoms
AMS-Qol - Quality of life questionnaire | Day 0
  Quality of life questionnaire to collect the level of difficulty experienced by the patient (from no problem to extreme problem) during the 4 weeks preceding the interview on activities such as : move; walk; maintain balance; talk; feed. It also assesses how the patient feels about his disease
AMS-Qol - Quality of life questionnaire | One year
  Quality of life questionnaire to collect the level of difficulty experienced by the patient (from no problem to extreme problem) during the 4 weeks preceding the interview on activities such as : move; walk; maintain balance; talk; feed. It also assesses how the patient feels about his disease
MOntreal Cognitive Assessment (Moca) score | Day 0
  Moca evaluates short-term memory, visual spatial skills, executive functions, attention, concentration, working memory, language, abstraction abilities, computing and orientation in time and space. Cognitive impairment is assessed on the score of 30 points (27-30: no cognitive impairment; 21-26: mild)
MOntreal Cognitive Assessment (Moca) score | One year
  Moca evaluates short-term memory, visual spatial skills, executive functions, attention, concentration, working memory, language, abstraction abilities, computing and orientation in time and space. Cognitive impairment is assessed on the score of 30 points (27-30: no cognitive impairment; 21-26: mild)
Brain MRI volume | Day 0
  Imaging data (severity and progression of putamen atrophy, bridge and cerebellum in mm3; magnitude and progression of white substance hypersignals on T2-FLAIR images in mm3
Brain MRI volume | One year
  Imaging data (severity and progression of putamen atrophy, bridge and cerebellum in mm3; magnitude and progression of white substance hypersignals on T2-FLAIR images in mm3

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France